CLINICAL TRIAL: NCT07292181
Title: Prevalence of Central Sensitization and Neuropathic Pain in Patients With Cervicogenic Headache: A Case-Control Study
Brief Title: Central Sensitization and Neuropathic Pain in Cervicogenic Headache
Status: Completed | Type: Observational
Sponsor: Gulseren Demir Karakilic (Other)
Responsible Party: Sponsor-Investigator, Gulseren Demir Karakilic, Assistant Professor, Principal Investigator, Bozok University
Organization: Bozok University (Other)
Other Study IDs: 2025-GOKAEK-2513_2025.07.02_50
Record Dates: First submitted 2025-12-05; First posted 2025-12-18 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Cervicogenic Headache; Central Sensitization; Neuropathic Pain
Keywords: Headache Disorders; Neck Pain; Pain Mechanisms; Psychological Distress; Sleep Quality; Quality of Life; Pain Assessment; Case-Control Study
MeSH Terms: conditions — Post-Traumatic Headache; Neuralgia; Headache Disorders; Neck Pain; Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patient group: Age range: 18 to 65 years Diagnosis of cervicogenic headache established according to the International Classification of Headache Disorders, 3rd edition criteria Recruited from outpatient clinics of Physical Medicine and Rehabilitation and Neurology Exclusion criteria: younger than 18 or older than 65, inability to communicate, illiteracy, refusal to participate, diabetes mellitus, hypothyroidism, chronic kidney disease, malignancy, neurological diseases associated with neuropathic pain, and rheumatic diseases such as rheumatoid arthritis, ankylosing spondylitis, or fibromyalgia
  Interventions: Other: Clinical assessment with standardized questionnaires
- Healthy Control Group: Age range: 18 to 65 years No diagnosis of cervicogenic headache or chronic pain conditions Age- and sex-matched to the patient group Voluntary participation Exclusion criteria: illiteracy, refusal to participate, diabetes mellitus, hypothyroidism, chronic kidney disease, malignancy, neurological diseases associated with neuropathic pain, and rheumatic diseases such as rheumatoid arthritis, ankylosing spondylitis, or fibromyalgia
  Interventions: Other: Clinical assessment with standardized questionnaires

INTERVENTIONS:
Other: Clinical assessment with standardized questionnaires — Participants in both the patient group and the healthy control group underwent a structured clinical assessment using validated instruments. The evaluation included measures of central sensitization, neuropathic pain features, headache-related disability, cervical functional impairment, psychological distress, sleep quality, and health-related quality of life. The instruments administered were the Central Sensitization Inventory, PainDETECT Questionnaire, Headache Impact Test, Neck Disability Index, Hospital Anxiety and Depression Scale, Jenkins Sleep Scale, and Short Form-36. No pharmacological or procedural intervention was applied as part of the study; the primary focus was on comparative assessment between groups.

SUMMARY:
Cervicogenic headache is a type of secondary headache that originates from the structures of the neck and can spread toward the head and facial regions. It is often one-sided and may be triggered by neck movement or sustained posture. The underlying mechanisms are thought to include abnormal processing of pain signals in the cervical spine and brainstem.

This case-control study was designed to examine whether individuals with cervicogenic headache show higher levels of central nervous system hypersensitivity and nerve-related pain compared with healthy individuals. The study also aimed to identify how these pain mechanisms are related to sleep, mood, and functional capacity.

The research was conducted at the Departments of Physical Medicine and Rehabilitation and Neurology of Yozgat Bozok University. Adults between 18 and 65 years of age who met the diagnostic criteria for cervicogenic headache were included. Age- and sex-matched healthy volunteers without chronic pain or neurological disorders were recruited as the control group.

Participants completed face-to-face interviews that included sociodemographic questions and a series of validated assessment tools measuring pain characteristics, psychological state, sleep quality, and quality of life. Ethical approval was obtained from the institutional review board, and all participants provided written informed consent prior to participation.

DETAILED DESCRIPTION:
Cervicogenic headache is a secondary headache that arises from disorders or dysfunctions of the cervical spine and its associated structures. Pain usually starts in the neck region and radiates toward the occipital and temporal areas. The condition can be provoked by neck movements and may be accompanied by neck stiffness or discomfort. The pathophysiology involves the convergence of sensory inputs from the cervical nerves and the trigeminal system at the brainstem level, which may lead to the referral of pain from the neck to the head.

In recent years, researchers have proposed that abnormal central nervous system activity and neuropathic pain components may contribute to the chronicity and treatment resistance of cervicogenic headache. Central hypersensitivity refers to increased excitability of pain-related neurons, while neuropathic pain is characterized by nerve dysfunction resulting in unusual pain sensations. A limited number of studies have addressed these mechanisms together in cervicogenic headache.

The present case-control study was conducted at Yozgat Bozok University to evaluate central nervous system hypersensitivity and neuropathic pain features in patients with cervicogenic headache compared to healthy controls. Data collection took place between July 2025 and October 2025. Individuals aged 18 to 65 years who fulfilled the diagnostic criteria for cervicogenic headache were included in the patient group. Exclusion criteria included neurological disorders, systemic diseases, cognitive impairment, or other rheumatic or chronic pain conditions. Healthy volunteers of similar age and sex without headache or chronic pain were selected as the control group.

Data were obtained using a structured questionnaire covering demographic and clinical information and a series of standardized scales. Pain-related disability was measured with the Headache Impact Test and the Neck Disability Index. Emotional status was evaluated with the Hospital Anxiety and Depression Scale. Sleep quality was assessed with the Jenkins Sleep Scale. Health-related quality of life was examined with the Short Form 36 questionnaire. The presence of nerve-related pain was assessed with the Pain Detect Questionnaire, and central nervous system hypersensitivity was evaluated with the Central Sensitization Inventory.

All assessments were administered face to face in the outpatient clinics by trained clinicians. Statistical analyses were performed using appropriate parametric and non-parametric tests after checking normality of data distribution. The study was approved by the Institutional Clinical Research Ethics Committee, and all participants signed written informed consent forms prior to enrollment.

ELIGIBILITY:
Eligibility Criteria

Inclusion Criteria:

* Adults aged 18 to 65 years
* Patient group: Clinical diagnosis of cervicogenic headache according to the International Classification of Headache Disorders, 3rd edition (ICHD-3) criteria
* Healthy control group: Age- and sex-matched individuals without cervicogenic headache or other chronic pain conditions
* Adequate cognitive function and literacy to complete questionnaires
* Voluntary participation with written informed consent

Exclusion Criteria:

* Age younger than 18 years or older than 65 years
* Inability to communicate effectively
* Illiteracy
* Refusal to participate
* Presence of systemic diseases including diabetes mellitus, hypothyroidism, chronic kidney disease, or malignancy
* Neurological diseases associated with neuropathic pain
* Rheumatologic diseases including rheumatoid arthritis, ankylosing spondylitis, or fibromyalgia
* Withdrawal of consent or incomplete data during the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population included 106 adult patients with cervicogenic headache and 106 age- and sex-matched healthy controls. Patients were recruited from outpatient clinics of Physical Medicine and Rehabilitation and Neurology at Bozok University, Turkey. Healthy volunteers were selected from the community and hospital staff who met the eligibility criteria.
Sampling Method: Non-Probability Sample
Enrollment: 72 (Actual)
Dates: Start 2025-07-03 (Actual); Primary Completion 2025-10-03 (Actual); Study Completion 2025-10-03 (Actual)

PRIMARY OUTCOMES:
Central Sensitization Inventory | At baseline
  Description: A 25-item self-report questionnaire that evaluates symptoms associated with central sensitization, including hypersensitivity, sleep disturbance, and emotional complaints.
  Scoring: Total score range 0-100. A score of 40 or higher suggests the presence of central sensitization.
  Turkish validation and reliability study: Conducted in 2021
PainDETECT Questionnaire | At baseline.
  Description: A self-administered screening tool for identifying neuropathic pain characteristics.
  Scoring: Total score range -1 to 38. Scores ≤12 indicate neuropathic pain is unlikely; scores ≥19 indicate neuropathic pain is likely; 13-18 indicates unclear classification.
  Turkish validation and reliability study: Conducted in 2013.

SECONDARY OUTCOMES:
Headache Impact Test (6 items) | At baseline
  Description: Measures the impact of headache on daily life, including pain severity, social functioning, and emotional well-being.
  Scoring: Total score range 36-78. Higher scores indicate greater impact. Severity cut-offs: ≤49 little or no impact; 50-55 some impact; 56-59 substantial impact; ≥60 severe impact.
  Turkish validation and reliability study: Conducted in 2021.
Neck Disability Index | At baseline
  Description: A 10-item questionnaire assessing how neck pain affects daily activities such as reading, working, and recreation.
  Scoring: Total score range 0-50, converted to percentage disability. Cut-off values: 0-4 no disability; 5-14 mild disability; 15-24 moderate disability; 25-34 severe disability; ≥35 complete disability.
  Turkish validation and reliability study: Conducted in 2009.
Hospital Anxiety and Depression Scale | At baseline
  Description: A 14-item scale with two subscales (7 for anxiety and 7 for depression).
  Scoring: Each subscale ranges 0-21. Higher scores reflect greater severity. Cut-offs: 0-7 normal, 8-10 borderline, ≥11 abnormal. Turkish validation and reliability study: Conducted in 1997.
Jenkins Sleep Scale | At baseline
  Description: A 4-item scale assessing sleep problems such as difficulty initiating or maintaining sleep and non-restorative sleep.
  Scoring: Total score range 0-20. Higher scores indicate poorer sleep quality. Turkish validation and reliability study: Conducted in 2018.
Short Form-36 Health Survey | At baseline
  Description: A 36-item instrument evaluating health-related quality of life across 8 domains: physical functioning, role limitations due to physical health, bodily pain, general health, vitality, social functioning, role limitations due to emotional problems, and mental health.
  Scoring: Each domain is scored 0-100, with higher scores indicating better quality of life.
  Turkish validation and reliability study: Conducted in 1999.

CONTACTS AND LOCATIONS:
Overall Officials: Gülseren Demir Karakılıç, Assistant Professor, Principal Investigator — Yozgat Bozok University
Locations (1):
- Yozgat Bozok University Faculty of Medicine, Department of Physical Medicine and Rehabilitation, Yozgat, Yozgat, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data (IPD) underlying the results reported in this study will be shared. Researchers can request access to de-identified data necessary to reproduce the study findings.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: IPD and supporting documents will be shared upon request following the publication of the study and will be available for up to 5 years.
Access Criteria: De-identified IPD and supporting documents will be provided to researchers who submit a methodologically sound research proposal. Requests should be made via email to the corresponding author and, once approved, data will be shared through a secure file transfer.
URL: https://hastane.bozok.edu.tr

REFERENCES:
- [Background] Kocyigit, H., Turkish validity and reliability of short-form 36. Drug Treat, 1999. 12: p. 102-106.
- [Background] Duruoz MT, Erdem D, Gencer K, Ulutatar F, Baklacioglu HS. Validity and reliability of the Turkish version of the Jenkins Sleep Scale in psoriatic arthritis. Rheumatol Int. 2018 Feb;38(2):261-265. doi: 10.1007/s00296-017-3911-2. Epub 2017 Dec 18. PMID 29250729
- [Background] Duzce Keles E, Birtane M, Ekuklu G, Kilincer C, Caliyurt O, Tastekin N, Is EE, Ketenci A, Neblett R. Validity and reliability of the Turkish version of the central sensitization inventory. Arch Rheumatol. 2021 Oct 18;36(4):518-526. doi: 10.46497/ArchRheumatol.2022.8665. eCollection 2021 Dec. PMID 35382371
- [Background] Alkan H, Ardic F, Erdogan C, Sahin F, Sarsan A, Findikoglu G. Turkish version of the painDETECT questionnaire in the assessment of neuropathic pain: a validity and reliability study. Pain Med. 2013 Dec;14(12):1933-43. doi: 10.1111/pme.12222. Epub 2013 Aug 7. PMID 23924395
- [Background] Aydemir, O., Hastane anksiyete ve depresyon olcegi Turkce formunun gecerlilik ve guvenilirligi. Turk Psikiyatri Derg., 1997. 8: p. 187-280.
- [Background] Telci EA, Karaduman A, Yakut Y, Aras B, Simsek IE, Yagli N. The cultural adaptation, reliability, and validity of neck disability index in patients with neck pain: a Turkish version study. Spine (Phila Pa 1976). 2009 Jul 15;34(16):1732-5. doi: 10.1097/BRS.0b013e3181ac9055. PMID 19770615
- [Background] Dikmen PY, Bozdag M, Gunes M, Kosak S, Tasdelen B, Uluduz D, Ozge A. Reliability and Validity of Turkish Version of Headache Impact Test (HIT-6) in Patients with Migraine. Noro Psikiyatr Ars. 2020 Apr 24;58(4):300-307. doi: 10.29399/npa.24956. eCollection 2021. PMID 34924791